CLINICAL TRIAL: NCT06377007
Title: Refractive Outcomes and Ocular Biometry of Two Swept-Source Optical Coherence Tomography-Based Biometers With Segmental or Equivalent Refractive Indices (ORION): A Non-Inferiority Randomized Clinical Trials
Brief Title: Refractive Outcomes and Ocular Biometry of Two Swept-Source Optical Coherence Tomography-Based Biometers With Segmental or Equivalent Refractive Indices (ORION)
Acronym: ORION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walailak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: WU66290; WU66290 (Other Grant/Funding Number: Walailak individual grant)
Record Dates: First submitted 2024-01-30; First posted 2024-04-22 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Biometry; SS-OCT; IOLMaster700; Argos
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IOLMaster 700 (Active Comparator): IOLMaster 700 represents the gold standard for measuring ocular biometry before cataract surgery, employing a single refractive index.
  Interventions: Device: IOLMaster 700 (Carl Zeiss Meditec AG)
- ARGOS (Experimental): ARGOS is a new device used to measure ocular biometry. It employs distinct refractive indices for different eye components such as the cornea, lens, and vitreous.
  Interventions: Device: Argos (Alcon Laboratories, Inc.)

INTERVENTIONS:
Device: IOLMaster 700 (Carl Zeiss Meditec AG) — Subjects will undergo measurements with the IOLMaster 700 device.
  Arms: IOLMaster 700
Device: Argos (Alcon Laboratories, Inc.) — Subjects will undergo measurements with the Argos device.
  Arms: ARGOS

SUMMARY:
Cataract surgery represents a common surgical intervention, encompassing the extraction of the opaque natural crystalline lens, followed by the substitution with an artificial intraocular lens (IOL). To ascertain an IOL possessing optimal power, antecedent to the surgery, preoperative evaluations are conducted through the utilization of a biometric devices. Diverse categories of these instruments are accessible, each harnessing distinct optical methodologies or mathematical algorithms to ascertain the most fitting IOL power. The principal objective of this study was to evaluate the ocular biometry and the predictive precision outcome of a biometer that uses standard keratometry to the prediction accuracy of another biometer that uses Total Keratometry.

DETAILED DESCRIPTION:
Two swept-source optical coherence tomography (SS-OCT) biometers, namely the Argos and the IOLMaster 700, will be employed for the preoperative assessment of the eyes of all subjects who will undergo cataract surgery at the Eye Outpatient Department (OPD) of Walailak University Hospital. The sequence of biometry measurements will be randomized among the subjects. In Group 1, measurements will be initially conducted using the Argos device, followed by the IOLMaster 700 device. Conversely, Group 2 subjects will undergo measurements with the IOLMaster 700 device first, followed by the Argos device. The sequence will be continuous without any breaks. The analysis will encompass the right eyes of each subject.

For the purpose of preoperative planning, the Argos device will utilize the Barrett Universal Formula II "K," whereas the IOLMaster 700 device will employ the Barrett Universal II TK formula. The objective for all eyes will be to achieve a plano outcome. In instances where the suggested intraocular lens (IOL) power differs between the two biometers, the IOL power recommended by the IOLMaster 700 device will be selected. Cataract surgeries will be exclusively performed by a seasoned surgeon (SM), who will adhere to a consistent approach involving a clear temporal incision (2.75 mm) followed by manual capsulorhexis. Refractive and visual outcomes will be evaluated within a postoperative timeframe of 28 to 42 days. Subjective refractions will be conducted by an optometrist, ensuring blinding to the biometry data.

The primary endpoint of this study will be the mean absolute prediction error exhibited by each SS-OCT biometer. The computation of the absolute prediction error will involve determining the absolute disparity between the predicted spherical equivalent refraction derived from preoperative planning and the actual measured spherical equivalent refraction (manifest). Secondary objectives will encompass the median absolute prediction error and the proportion of eyes with an absolute prediction error equal to or less than 0.25 D and 0.5 D.

ELIGIBILITY:
Inclusion Criteria:

• Patients with cataract and/or presbyopia who will undergo intraocular lens implantation.

Exclusion Criteria:

* Central corneal thickness less than 490 mm or greater than 600 mm
* Contact lens use within 2 months of cataract surgery
* Severe dry eye
* Corneal or retinal disease affecting visual outcome
* Corneal astigmatism greater than 1.00 D
* Prior corneal refractive surgery
* Dense cataract that does not allow measurements to be taken with an optical biometrics system.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean absolute prediction error | 4 weeks
  Mean absolute prediction error determining by the absolute disparity between the predicted spherical equivalent refraction derived from preoperative planning and the actual measured spherical equivalent refraction (manifest) from both devices (IOLMaster 700 and Argos)

SECONDARY OUTCOMES:
Proportion of eyes with an absolute prediction error equal to or less than 0.25 | 4 weeks
  The proportion of eyes with an absolute prediction error equal to or less than 0.25 D and 0.5 D.

CONTACTS AND LOCATIONS:
Locations (1):
- Walailak University, Nakhon Si Thammarat, Thailand